CLINICAL TRIAL: NCT01514994
Title: Treatment of Critical Aortic Valve Stenosis Using a Novel Valvuloplasty Scoring Balloon Catheter: a First-in-Man Study
Brief Title: Valvuloplasty Scoring Balloon Catheter First-in-Man Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Spectranetics Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ST-1486
Record Dates: First submitted 2012-01-11; First posted 2012-01-23 (Estimated); Last update posted 2016-04-18 (Estimated); Status verified 2016-04

CONDITIONS: Aortic Valve Stenosis
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- AngioScore's Valvuloplasty Scoring Balloon (Experimental)
  Interventions: Device: AngioScore's Valvuloplasty Scoring Balloon

INTERVENTIONS:
Device: AngioScore's Valvuloplasty Scoring Balloon — All patients will receive treatment for their aortic valve stenosis with the Valvuloplasty Scoring Balloon Catheter.

SUMMARY:
The Valvuloplasty Scoring Balloon First-in-Man study is a prospective, single arm, two phase, observational registry to demonstrate the safety and efficacy of the Valvuloplasty Scoring Balloon Catheter for the treatment of critical aortic valve stenosis.

DETAILED DESCRIPTION:
Phase 1 will enroll patient who are scheduled to undergo open surgical aortic valve replacement and will have the Valvuloplasty Scoring Balloon delivered to their stenotic aortic valve through a standard aortotomy and deployed immediately prior to valve replacement.

Phase 2 will enroll patients with aortic valve stenosis who are deemed to not be suitable candidates for elective surgical aortic valve replacement and in whom the investigational Valvuloplasty Scoring Balloon will be used as a stand-alone Valvuloplasty procedure or "bridge" to trans-catheter aortic valve implantation (TAVI) or surgery.

ELIGIBILITY:
Inclusion Criteria:

* Native, degenerative-calcific, tricuspid, aortic valve stenosis with echocardiographic derived criteria: mean gradient of >40 mm Hg or Doppler peak systolic velocity greater than 4.0 m/s or an initial aortic valve area < 0.8 cm2.
* Symptomatic aortic valve disease as demonstrated by CCS Functional Class II or greater
* Aortic valve annulus of greater than or equal to 18 mm and less than or equal to 28 mm measured on pre-procedure TTE.
* Phase 1 patients must be scheduled for a surgical aortic valve replacement.
* Phase 2 patients must not be suitable candidates for elective surgical aortic valve replacement.

Exclusion Criteria:

* Recent myocardial infarction (<30days)
* Unicuspid or bicuspid aortic valve or non-calcific aortic valve stenosis
* Any sepsis, including active endocarditis
* Concomitant 2+ or greater aortic valve valve regurgitation
* LVEF < 20%
* CVA or TIA within the previous 6 months
* Previous aortic valve replacement (bioprosthetic or mechanical)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2012-06; Primary Completion 2014-12 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Procedural Success | 1 day
  Procedural success defined as a >50% increase in the aortic valve effective orifice area and less than or equal to 2+ valvular regurgitation at the end of the percutaneous valvuloplasty procedure utilizing echocardiography, hemodynamic measurements and angiography.
Number of participants who do not experience death, stroke, myocardial infarction or emergency cardiac surgery during their hospitalization. | Participants will be followed for the duration of the hospital stay, an expected average of 48 hours
  Freedom from in-hospital death, stroke, myocardial infarction or emergency cardiac surgery

CONTACTS AND LOCATIONS:
Overall Officials: John G. Webb, MD, Principal Investigator — St. Paul's Hospital, Vancouver, Canada
Locations (1):
- St. Paul's Hospital, Vancouver, British Columbia, Canada